CLINICAL TRIAL: NCT02167100
Title: Patient Retention in HIV Medical Care in a Primary Care Practice in Australia
Acronym: RiC
Status: Completed | Type: Observational
Sponsor: Holdsworth House Medical Practice (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Dr. Mark Bloch, Director, Holdsworth House Medical Practice
Other Study IDs: Retention in Care Audit; HIV Retention in Care (Other: HHMP)
Record Dates: First submitted 2014-06-05; First posted 2014-06-18 (Estimated); Last update posted 2015-09-21 (Estimated); Status verified 2015-09

CONDITIONS: HIV
Keywords: HIV; Highly Active Antiretroviral Therapy; Patient Care; Patient Care Management; Lost to Follow-Up

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Retained in Care: Each patient who had at least 2 practice visits separated by ≥90 days in a year involving HIV laboratory monitoring until 31st of March 2014.
- Lost to follow-up (LTFU): Each patient who had at 2 practice visits separated by ≥90 days in a year involving HIV laboratory monitoring but did not maintain regular attendance at HHMP until 31st March, 2014.

SUMMARY:
The purpose of this study is to determine linkage and retention in care in patients with HIV infection and reasons for loss to follow up Care in a High HIV-caseload Inner City Primary Care Practice in Sydney, Australia.

The investigators hypothesise that patients attending HHMP will have higher rates of linkage and retention in care than the US HIV-infected population, and equivalent to Australian modelling.

DETAILED DESCRIPTION:
Many deficits in the spectrum of engagement in HIV care are still present and pose barriers to optimal treatment outcomes. These deficits include late diagnosis of HIV , insufficient linkage to and retention in care (RiC), poor usage of antiretroviral therapy (ART), and suboptimal adherence to ART. Based on data from the United States Center for Disease Control, where a cascade of care has been developed examining total numbers with HIV, numbers diagnosed, numbers linked to care, numbers on treatment and numbers on effective treatment; only about a quarter of persons living with HIV (PLWH) in the US are effectively in care, with undetectable HIV viral load.

Current data available in an Australian population are based on a patient modelling analysis, highlighting the lack of real cohort data from clinical practices managing HIV patients in Australia.

Appropriate continuum in care is relevant both for the prognosis of the single patient and for reducing the HIV transmission in the community. Substance use, high CD4 cell counts and young age seem to be risk factors for failure to establish care.

Holdsworth House Medical Practice (HHMP) is a high HIV-caseload community medical practice in inner city Sydney that provides a Continuum of Care for HIV-infected patients, from counselling and testing to antiretroviral treatment.

In this audit, we will examine retrospectively the case notes of >2000 HIV-infected patients who attended HHMP in Darlinghurst, Sydney, New South Wales with documented HIV infection from 1st January 2009 to 31st March 2014.

The primary objective of this audit is to determine linkage and retention in care in patients with HIV-1 infection and reasons for loss to follow up. Audit findings will be systematically evaluated, and where indicated, changes will be made with the aim of monitoring linkage and retention in care.

The initial audit will include patients with documented HIV-1 infection, who have attended the practice over a 5-year period (2009 - 2014) for at least 2 visits that are separated by 3 - 12 months, with specific laboratory tests (i.e. CD4 T lymphocyte count, plasma HIV RNA etc.) performed either on-site or at a co-management site.

Retention in care will be assessed by the number of visits to either HHMP or co-management sites over a 5-year period (2009 - 2014) for each patient audited. Demographic data along with laboratory test results and antiretroviral therapy regime data will be collected to assess factors associated with retention in care.

ELIGIBILITY:
Inclusion Criteria:

* Documented HIV-1 infection
* Attendance during the study period for at least 2 visits >3 months and <12 months apart with measured laboratory virological or immunological markers (either on-site or at a co-management site)

Exclusion Criteria:

* Attendance by patient with HIV infection who does not have laboratory markers of HIV viral load or CD4 count measured
* Incomplete/inaccessible patient records to enable patient to meet inclusion criteria
* Initial visit after 1st January 2014

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV-infected patients attending HHMP from 1st January 2009 to 31st March 2014 inclusive, who had at least 2 practice visits separated by ≥90 days in a year involving HIV laboratory monitoring whilst attending HHMP.
Sampling Method: Non-Probability Sample
Enrollment: 1537 (Actual)
Dates: Start 2014-06; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
The primary outcome measures are the rates of current linkage and retention in care for HIV-infected adults at Holdsworth House Medical Practice (HHMP) over a 5-year period | Up to 5 years

SECONDARY OUTCOMES:
A secondary outcome measure is to determine the factors associated with loss to follow up (LTFU) in the study population over a 5-year period | Up to 5 years

OTHER OUTCOMES:
Determining the reasons for LTFU - death, move to another practice, move interstate or overseas, other reason, unknown | Up to 5 years
The proportion of patients on antiretroviral therapy vs. not on therapy | Up to 5 years
The proportion of patients with undetectable viral load i.e. most recent plasma HIV RNA <50 copies/mL | Up to 5 years
The proportion of patients with normal immunity i.e. most recent CD4 >500 cells/μL | Up to 5 years
The proportion of treatment-naïve patients with CD4>500 cells/μL. | Up to 5 years
Antiretroviral regimen (including single-tablet-regimen) association with retention in care and LTFU | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Mark T Bloch, MBBS, Principal Investigator — Holdsworth House Medical Practice
Locations (1):
- Holdsworth House Medical Practice, Darlinghurst, New South Wales, Australia

REFERENCES:
- [Background] Hall HI, Halverson J, Wilson DP, Suligoi B, Diez M, Le Vu S, Tang T, McDonald A, Camoni L, Semaille C, Archibald C. Late diagnosis and entry to care after diagnosis of human immunodeficiency virus infection: a country comparison. PLoS One. 2013 Nov 5;8(11):e77763. doi: 10.1371/journal.pone.0077763. eCollection 2013. PMID 24223724
- [Background] Gardner EM, McLees MP, Steiner JF, Del Rio C, Burman WJ. The spectrum of engagement in HIV care and its relevance to test-and-treat strategies for prevention of HIV infection. Clin Infect Dis. 2011 Mar 15;52(6):793-800. doi: 10.1093/cid/ciq243. PMID 21367734
- [Background] Centers for Disease Control and Prevention (CDC). Vital signs: HIV prevention through care and treatment--United States. MMWR Morb Mortal Wkly Rep. 2011 Dec 2;60(47):1618-23. PMID 22129997
- [Background] Mugavero MJ, Lin HY, Willig JH, Westfall AO, Ulett KB, Routman JS, Abroms S, Raper JL, Saag MS, Allison JJ. Missed visits and mortality among patients establishing initial outpatient HIV treatment. Clin Infect Dis. 2009 Jan 15;48(2):248-56. doi: 10.1086/595705. PMID 19072715
- [Background] Das M, Chu PL, Santos GM, Scheer S, Vittinghoff E, McFarland W, Colfax GN. Decreases in community viral load are accompanied by reductions in new HIV infections in San Francisco. PLoS One. 2010 Jun 10;5(6):e11068. doi: 10.1371/journal.pone.0011068. PMID 20548786
- [Background] Fang CT, Hsu HM, Twu SJ, Chen MY, Chang YY, Hwang JS, Wang JD, Chuang CY; Division of AIDS and STD, Center for Disease Control, Department of Health, Executive Yuan. Decreased HIV transmission after a policy of providing free access to highly active antiretroviral therapy in Taiwan. J Infect Dis. 2004 Sep 1;190(5):879-85. doi: 10.1086/422601. Epub 2004 Jul 22. PMID 15295691
- [Background] Giordano TP, Visnegarwala F, White AC Jr, Troisi CL, Frankowski RF, Hartman CM, Grimes RM. Patients referred to an urban HIV clinic frequently fail to establish care: factors predicting failure. AIDS Care. 2005 Aug;17(6):773-83. doi: 10.1080/09540120412331336652. PMID 16036264